CLINICAL TRIAL: NCT01531647
Title: A Study to Evaluate the Potential Drug-Drug Interaction Between Danoprevir/Low-Dose Ritonavir When Given With Raltegravir in Healthy Adult Volunteers
Brief Title: A Study of Drug-Drug Interaction Between Danoprevir/Low-Dose Ritonavir and Raltegravir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: NP28088
Record Dates: First submitted 2012-01-19; First posted 2012-02-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Raltegravir Potassium; Ritonavir

ARMS (2):
- Period 1 Control (Active Comparator)
  Interventions: Drug: raltegravir
- Period 2 danoprevir/ritonavir (Experimental)
  Interventions: Drug: danoprevir; Drug: raltegravir; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — 100 mg q12h Days 8-21
  Arms: Period 2 danoprevir/ritonavir
Drug: raltegravir — 400 mg q12h Days 1-4 and 18-21
Drug: ritonavir — 100 mg q12h Days 8-21
  Arms: Period 2 danoprevir/ritonavir

SUMMARY:
This open-label, multiple dose, single sequence crossover study will evaluate the drug-drug interaction between danoprevir/low-dose ritonavir and raltegravir in healthy volunteers. Subjects will receive raltegravir on Days 1-4 and, after a washout period of 3 days, danoprevir and low-dose ritonavir on Days 8-21, in combination with raltegravir on Days 18-21.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male and female adults, 18 - 55 years of age, inclusive
* Healthy status defined by absence of evidence of any active or chronic disease
* Medical history without major, recent, or ongoing pathology
* Weight >/= 50.0 kg
* Body mass index (BMI) 18.0 - 32-0 kg/m2
* Willingness to abstain from alcohol, xanthine-containing beverages or food (e.g. coffee, tea, cola, chocolate, "energy drinks") from 48 hours prior to entry in the clinical site until discharge
* Females of child-bearing potential and males and their female partners of child-bearing potential must agree to use 2 forms of contraception, one of which must be a barrier method, during the study and for 90 days after the last drug administration. Acceptable barrier forms of contraception are condom and diaphragm; acceptable non-barrier forms of contraception for this study are non-hormonal intrauterine device (IUD) and/or spermicide

Exclusion Criteria:

* Pregnant or lactating females or males with female partners who are pregnant or lactating
* Any history of clinically significant cardiovascular or cerebrovascular disease, hypertension, and/or infections
* Positive test for drugs of abuse at screening or prior to admission to the clinical site during any study period
* Positive for hepatitis B, hepatitis C or HIV infection
* Current smokers or subjects who have discontinued smoking less than 6 months prior to first dose of study medication
* Use of hormonal contraceptives within 30 days before the first dose of study medication
* History of clinically significant drug-related allergy (such as anaphylaxis) or hepatotoxicity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Effect of steady-state ritonavir-boosted danoprevir on steady-state raltegravir pharmacokinetics: Area under the concentration-time curve (AUC) | approximately 2 months

SECONDARY OUTCOMES:
Effect of steady-state raltegravir on danoprevir/ritonavir pharmacokinetics: Area under the concentration-time curve (AUC) | Pre-dose Days 8. 14, 15, 16 and 20, pre-and up to 24 h post-dose Days 17 and 21
Safety: Incidence of adverse events | approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States